CLINICAL TRIAL: NCT01760824
Title: Ten Days Quadruple Versus Sequential Therapy as Empirical First and Second Line Treatment for Helicobacter Pylori Eradication: a Randomized Crossover Trial
Brief Title: Quadruple Versus Sequential Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW 11-221
Record Dates: First submitted 2012-12-29; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Sequential; Quadruple; First; Line; Helicobacter; pylori; infection
MeSH Terms: conditions — Infections | interventions — Esomeprazole; BID protein, human; Amoxicillin; Clarithromycin; Metronidazole; bismuth tripotassium dicitrate; Tetracycline; Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequential therapy (Experimental): Esomeprazole 20mg bid for 10 days, amoxicillin 1g bid for first 5 days, clarithromycin 500mg bid for last 5 days and metronidazole 400mg qid for last 5 days
  Interventions: Drug: Sequential therapy; Drug: Quadruple therapy
- Quadruple therapy (Active Comparator): Esomeprazole 20mg bid, metronidazole 400mg aid, bismuth sub citrate 120mg aid and tetracycline 500mg qid, all for 10 days
  Interventions: Drug: Sequential therapy; Drug: Quadruple therapy

INTERVENTIONS:
Drug: Sequential therapy — Esomeprazole 20mg bid for 10 days, amoxicillin 1g bid for first 5 days, clarithromycin 500mg bid for last 5 days and metronidazole 400mg qid for last 5 days
  Other Names: Esomeprazole (Nexium) 20mg bid for 10 days; Amoxicillin 1g bid for first 5 days; Clarithromycin (Klacid) 500mg bid for last 5 days; Metronidazole (Flagyl) 400mg qid for last 5 days
Drug: Quadruple therapy — Esomeprazole 20mg bid, metronidazole 400mg qid, bismuth sub citrate 120mg qid and tetracycline 500mg qid, all for 10 days
  Other Names: Esomeprazole (Nexium) 20mg bid; Metronidazole (Flagyl) 400mg qid; Bismuth subcitrate 120mg qid; Tetracycline 500mg qid; all for 10 days

SUMMARY:
Helicobacter pylori (HP), a bacterium present in many people's stomachs, is one of the major causes of ulcers and cancers. Up to 20% of patients infected with H. pylori may develop peptic ulcers. However, failure rate is rising due to multiple resistant H. pylori infection. The eradication rate of first line clarithromycin based therapy has fallen to below 80%. Both quadruple and sequential treatment regime has been proposed as the first-line empirical regime. Nevertheless, comparison in terms of efficacy and side effects between the two regime remained unknown. The aim of this clinical trial is to compare the efficacy and tolerability of H. pylori eradication with a 10-day quadruple therapy versus sequential therapy as empirical first and second line treatment.

DETAILED DESCRIPTION:
Helicobacter pylori (HP), a bacterium present in many people's stomachs, is one of the major causes of ulcers and cancers. Up to 20% of patients infected with HP may develop peptic ulcers. However, failure rate is rising due to multiple resistant HP infection. The eradication rate of first line clarithromycin based therapy has fell to below 80% and increasing number of patients also failed the second line quadruple therapy. The aim of this clinical trial is to compare the efficacy and tolerability of H. pylori eradication with a 10-day quadruple therapy versus sequential therapy as empirical first and second line treatment.

Methods: Eligible H. pylori positive patients were randomized to receive either QUAD (esomeprazole 20mg twice daily, bismuth subcitrate 120mg four times daily, tetracycline 500mg four times daily and metronidazole 400mg four times daily) for 10 days or SEQ (esomeprazole 20mg twice daily for 10 days, amoxicillin 1g twice daily for first 5 days, clarithromycin 500mg twice daily and metronidazole 400mg four time daily for the subsequent 5 days). All patients returned 8 weeks after completing the treatment for a Urea Breath Test (UBT) to confirm eradication. Patients who failed their respective therapy were crossover to receive the alternative regimen.

ELIGIBILITY:
Inclusion Criteria:

* patients with age 18 or above, diagnosed to have gastric HP infection

Exclusion Criteria:

* Patients with age less than 18, with past allergy to the study medications, concurrent critical illnesses, a history of previous upper gastrointestinal surgery, intake of nonsteroidal anti-inflammatory drugs, antibiotics, probiotics, bismuth preparation, proton pump inhibitors, anticoagulants or steroids in the previous one month, pregnant or breast-feeding women, drug abusers or alcoholic, history of previous H. Pylori treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 8 weeks after treatment
  Percentage of patients successfully eradicated Helicobacter pylori infection confirmed by urea breath test

SECONDARY OUTCOMES:
Development of side effects | 10 days
  Patients to document side effects during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong SAR, Hong Kong

REFERENCES:
- [Derived] Liu KS, Hung IF, Seto WK, Tong T, Hsu AS, Lam FY, But DY, Wong SY, Leung WK. Ten day sequential versus 10 day modified bismuth quadruple therapy as empirical firstline and secondline treatment for Helicobacter pylori in Chinese patients: an open label, randomised, crossover trial. Gut. 2014 Sep;63(9):1410-5. doi: 10.1136/gutjnl-2013-306120. Epub 2013 Dec 2. PMID 24295850